CLINICAL TRIAL: NCT06041685
Title: Effect of Local Warming for Arterial Catheterization in Pediatric Cardiac Surgery: A Prospective Randomized Controlled Study
Brief Title: Effect of Local Warming for Arterial Catheterization in Pediatric Anesthesia
Acronym: WARM-PA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Fund assistant professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05-2023-183
Record Dates: First submitted 2023-09-08; First posted 2023-09-18 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-warming group (C) (No Intervention): After induction, the baseline artery ultrasonography images are collected for the internal diameter and cross-sectional area of the artery. In the non-warming group (C), local warming is not applied on the catheterization site. Before catheterization, the artery ultrasonography images are collected. Then, arterial catheterization is applied.
- Warming group (W) (Experimental): In the warming group (W), local warming is applied on the catheterization site. Before catheterization, the artery ultrasonography images are collected. Then, arterial catheterization is done.
  Interventions: Procedure: local warming

INTERVENTIONS:
Procedure: local warming — local warming on the site for arterial catheterization using forced air warmer
  Arms: Warming group (W)

SUMMARY:
The increase in internal diameter (ID) and cross-sectional area (CSA) may facilitate better arterial catheterization. Since an increase in body temperature can cause peripheral vasodilation, we aimed to determine if local warming of the radial artery (RA) catheterization site could improve the success rate of catheterization in pediatric patients.

DETAILED DESCRIPTION:
This randomized, controlled study enrolls 126 pediatric patients aged ≤ 2 years who were scheduled for heart surgery. They are randomized into non-warming (C) and warming (W) groups. After induction, the baseline artery ultrasonography images are collected. In the warming group (W), local warming is applied on the catheterization site. Before catheterization, the artery ultrasonography images are collected. The primary outcome is the first-attempt success rate. The secondary outcomes included the ID and CSA of the artery and overall complications.

ELIGIBILITY:
Inclusion Criteria:

* aged ≤ 2 years
* cardiac surgery with peripheral artery catheterization

Exclusion Criteria:

* unstable vital signs
* pre-existing arterial catheter (exception of umbilical artery catheterization)

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
first-attempt success rate of arterial catheterization | baseline, imediate after arterial catheterization
  The first-attempt success rate of pediatric peripheral arterial catheterization in the non-warming group, or warming group

SECONDARY OUTCOMES:
internal diameter (ID) and cross-sectional area (CSA) | baseline, imediate after arterial catheterization in the non-warming group, or warming group
  internal diameter (ID) and cross-sectional area (CSA)

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, Principal Investigator — Pusan National University
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christen S, Delachaux A, Dischl B, Golay S, Liaudet L, Feihl F, Waeber B. Dose-dependent vasodilatory effects of acetylcholine and local warming on skin microcirculation. J Cardiovasc Pharmacol. 2004 Dec;44(6):659-64. doi: 10.1097/00005344-200412000-00006. PMID 15550784
- [Background] Al-Hakim R, Hedge JC, Jahangiri Y, Kaufman JA, Galuppo R, Farsad K. Palmar Warming for Radial Artery Vasodilation to Facilitate Transradial Access: A Randomized Controlled Trial. J Vasc Interv Radiol. 2019 Mar;30(3):421-424. doi: 10.1016/j.jvir.2018.10.021. PMID 30819486
- [Background] Barcroft H, Edholm OG. The effect of temperature on blood flow and deep temperature in the human forearm. J Physiol. 1943 Jun 30;102(1):5-20. doi: 10.1113/jphysiol.1943.sp004009. No abstract available. PMID 16991588